CLINICAL TRIAL: NCT04272840
Title: Adapting a National Glycemic Index Education Platform for Nova Scotian Patients and Clinicians Treating Gestational Diabetes Mellitus Using Distance Education Strategies.
Brief Title: The Impact of Glycemic Index Education on Lowering Dietary GI in Gestational Diabetes Mellitus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IWK Health Centre (Other)
Collaborators: Mount Saint Vincent University (Other); Dalhousie University (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Shannan Grant, Affiliated Scientist, IWK Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI in GDM Online
Record Dates: First submitted 2019-10-20; First posted 2020-02-17 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Gestational Diabetes; Glycaemic or Glycemic Index; Nutrition; Education; Behaviour
MeSH Terms: conditions — Diabetes, Gestational; Behavior

STUDY DESIGN:
Intervention Model Description: Prospective Randomized Control Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Participants will attend a 30-45 min workshop. Trainees will review Diabetes Canada Clinical Practice Guidelines Job Aids (Just the Basics, the Handy Portion Guide, and Basic Carbohydrate Counting) and teach data provision skills (how to complete a three day diet record).
- Low Glycemic Index (Experimental): Standard care + Glycemic Index. Participants will attend a 30-45 min workshop. Trainees will review Diabetes Canada Clinical Practice Guidelines Job Aids (Just the Basics, the Handy Portion Guide, and Basic Carbohydrate Counting) and teach data provision skills (how to complete a three day diet record). Diabetes Canada and Dietitian's Canada resources on glycemic index will also be reviewed: the Glycemic Index Food Guide, Flip Cards, and Recipes.
  Interventions: Behavioral: Low Glycemic Index Education

INTERVENTIONS:
Behavioral: Low Glycemic Index Education — Educational materials layering Glycemic Index education onto Canada's Food Guide and Diabetes Canada recommendations.
  Arms: Low Glycemic Index

SUMMARY:
Gestational Diabetes Mellitus (GDM) incidence is increasing worldwide, and within Canada, the Atlantic provinces statistically have been found to have highest prevalence of diabetes. Increasing evidence supports the benefit of following a low glycaemic index (GI) diet in GDM and the Canadian Diabetes Guidelines recommends replacing high GI foods for low GI foods. Despite recommendation to adapt a low GI diet in GDM, there are limitations and barriers recognized to GI utility largely focused on knowledge translation. There is sufficient research to support a low GI diet in benefiting outcomes of GDM, therefore the GI in GDM Online trial will investigate the feasibility and effectiveness of a distance low GI education intervention, adapted from Diabetes Canada's GI materials, on producing a difference in average dietary GI between a group with the intervention and standard care.

DETAILED DESCRIPTION:
The incidence of Gestational Diabetes Mellitus (GDM) has been progressively increasing worldwide, with a global prevalence of gestational hyperglycaemia estimated at 16.9%. In Canada, Atlantic provinces have been recorded with the highest prevalence of diabetes at 6%. The Diabetes Canada Practice Guidelines recommends the low glycemic index (GI) diet to type 1 and 2 diabetes mellitus and has recently updated its guidelines to include a recommendation for GDM. This said, barriers to GI knowledge translation have been identified. This study uses a prospective parallel randomized control trial design. Procedures and materials have been adapted from NCT01589757. The Kirkpatrick Model (Reaction, Learning, Behaviour, and Results) informed intervention development and evaluation strategies. The purpose of this study is to evaluate whether a distance low GI education intervention, adapted from Diabetes Canada's GI education materials, will significantly yield a lower average GI (primary outcome) in participants than traditional standard care medical nutrition therapy for Gestational Diabetes Mellitus. We hypothesize that participants who receive the low GI intervention will have a lower dietary GI than those who received usual IWK standard care for GDM.

ELIGIBILITY:
Inclusion Criteria:

* Of or over 18 years of age
* Diagnosed with GDM according to Diabetes Canada
* At or over than 20 weeks gestation
* At or less than 32 weeks gestation
* Being followed at IWK Health Centre
* Willing and able to give informed consent
* Willing and able to complete study protocol
* Currently living in Nova Scotia

Exclusion Criteria; women who:

* have been diagnosed with acute or chronic illness, other than GDM and PCOS, that may impact carbohydrate digestion metabolism.
* are currently taking a medication (other than insulin) that may affect carbohydrate metabolism.
* have multi-fetal pregnancy in current pregnancy.
* have insurmountable language barriers.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
Transfer/KM Level 3: Change in average dietary GI | From baseline to 4-6 weeks postpartum
  Average dietary GI; diet record at baseline, 4-6 weeks post-intervention, 4-6 weeks postpartum

SECONDARY OUTCOMES:
Satisfaction/ KM Level 1: Reaction | From baseline to 4-6 weeks postpartum
  Mixed form Questionnaire (GIQ): Close ended format with True or False, Multiple Choice, and Likert Scale choices. Open-ended questions for feedback.
Knowledge/KM Level 2: Learning | From baseline to 4-6 weeks postpartum
  Average Quiz Score: Close-ended format, Scored by correct answers.
Acceptability and Applicability of Education/KM Level 3: Transfer (Behaviour Change) | From 4-6 weeks post-intervention to 4-6 weeks post-partum
  Mixed form Questionnaire (GIQ): Close ended format using Likert Scale and True or False choices. Open-ended questions for feedback.
Results/KM Level 4: Glycemic Control (rate of Self-monitored blood glucose levels within range) | From Baseline to 4-6 weeks post-partum
  Medical Record (standard care 2-4 time-points per day)
Maternal Demographics (eg. age, ethnicity, language spoken, education level and work status) | Baseline
  Mixed-form Questionnaire (GIQ) and Medical Chart
Maternal Height | Baseline
  Medical Record, measured in cm.
Maternal Pre-Pregnancy body weight | Baseline
  Medical Record, measured in kg.
Maternal Weight, during pregnancy | From Baseline to 4-6 weeks post-partum.
  Medical Record, measured in kg.

CONTACTS AND LOCATIONS:
Overall Officials: Shannan Grant, PhD, PDt, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diabetes Canada Clinical Practice Guidelines Expert Committee; Feig DS, Berger H, Donovan L, Godbout A, Kader T, Keely E, Sanghera R. Diabetes and Pregnancy. Can J Diabetes. 2018 Apr;42 Suppl 1:S255-S282. doi: 10.1016/j.jcjd.2017.10.038. No abstract available. PMID 29650105
- [Background] Draffin CR, Alderdice FA, McCance DR, Maresh M, Harper Md Consultant Physician R, McSorley O, Holmes VA. Exploring the needs, concerns and knowledge of women diagnosed with gestational diabetes: A qualitative study. Midwifery. 2016 Sep;40:141-7. doi: 10.1016/j.midw.2016.06.019. Epub 2016 Jun 29. PMID 27553869
- [Background] Layes, A. The Burden of Diabetes in Atlantic Canada. Public Health Agency of Canada, Atlantic Regional Office; 2011.
- [Background] Grant SM, Wolever TMS. Perceived barriers to application of glycaemic index: valid concerns or lost in translation? Nutrients. 2011 Mar;3(3):330-340. doi: 10.3390/nu3030330. Epub 2011 Feb 28. PMID 22254100
- [Background] Johnston S, Coyer FM, Nash R. Kirkpatrick's Evaluation of Simulation and Debriefing in Health Care Education: A Systematic Review. J Nurs Educ. 2018 Jul 1;57(7):393-398. doi: 10.3928/01484834-20180618-03. PMID 29958308
- See also: Statistics Canada: Diabetes (2017) — https://www150.statcan.gc.ca/n1/pub/82-625-x/2018001/article/54982-eng.pdf